CLINICAL TRIAL: NCT05855525
Title: Real-time fMRI for Insular Cortex Brain State-triggered Experience Sampling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2208009393; 1R21MH129630-01A1 (NIH)
Record Dates: First submitted 2023-03-30; First posted 2023-05-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real-time fMRI (Experimental): Participants will repeatedly and intermittently report the content of their ongoing, self-generated experiences based on an experience-sampling protocol in which self-report ratings will be triggered based on real-time analysis of the participant's current brain state. The protocol will be conducted while participants are undergoing MRI scanning.
  Interventions: Behavioral: Experience sampling

INTERVENTIONS:
Behavioral: Experience sampling — Participants will repeatedly and intermittently report the content of their ongoing, self-generated experiences based on an experience-sampling protocol in which self-report ratings will be triggered based on real-time analysis of the participant's current brain state. The protocol will be conducted while participants are undergoing MRI scanning.

SUMMARY:
In a neuroimaging session, study participants will repeatedly and intermittently report the content of their ongoing, self-generated experiences based on an experience-sampling protocol in which self-report ratings will be triggered based on real-time analysis of the participant's current brain state. The protocol will be conducted while participants are undergoing MRI scanning.

DETAILED DESCRIPTION:
The investigators will develop a new approach called real-time functional MRI (fMRI)-triggered experience-sampling to efficiently sample spontaneous neural events (of a predefined type) and to map those events to specific qualities of self-generated experiences. Within 60 healthy adults, the investigators will use online (real-time) fMRI analysis to detect brain activations and trigger the appearance of visual rating scales so that participants can report their experiences immediately after the occurrence of a neural event of interest. The investigators will develop and validate the approach with a focus on real-time fMRI analysis of the dorsal anterior insular cortex (daIC), a brain region implicated in salience detection that is consistently identified as having aberrant structure, function, and connectivity in psychiatric illness at a transdiagnostic level. Aim 1 is to determine whether spontaneous daIC activation events are time-locked to instances of salient, high-arousal self-generated experience. The investigators will sample self-generated experiences both during instances of daIC activation and during baseline (intermediate daIC activity) events. The investigators hypothesize that daIC activation, relative to baseline events, will be time-locked to self-generated experiences with higher subjective ratings of arousal and vividness (regardless of affective valence). Aim 2 is to determine how distinct instances of daIC activation are coupled to physiological and whole-brain activity. Using a hypothesis-driven approach, the investigators will determine whether spontaneous fMRI activations in the daIC are associated with pupil dilation and activation of the locus coeruleus, a subcortical generator of arousal-related neuromodulation. Additionally, using a more data-driven approach, the investigators will test whether different instances of daIC activation are associated with multiple, distinct whole-brain co-activation patterns, and whether these co-activation patterns are associated with fluctuations in subjective affect (positive vs. negative experiences). If successful, the protocols can later be applied in patients with psychiatric illness and to potentially guide the development of interventions (e.g., neurostimulation, neurofeedback) that aim to target the neural processes that produce self-generated experiences that are core to mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35

Exclusion Criteria:

* History of psychiatric or neurological disorder
* contraindication for MRI

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants showing an association between self-reported arousal (simple rating scale) and fMRI activation level in anterior insula | Two sessions over one month
  Participants will rate their subject arousal level on trials that are triggered by anterior insula activation (using real-time fMRI analysis) and control trials not involving anterior insula activation. The outcome is the number of participants showing an association between self-reported arousal and fMRI activation in anterior insula.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Kucyi, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data generated from this study will become publicly available. After de-identifying and anonymizing all neuroimaging and behavioral data, the investigators plan to share data via the National Institute of Mental Health Data Archive.
Supporting Information: Study Protocol
Time Frame: Availability: December 2024 until 2030
Access Criteria: Publicly available